CLINICAL TRIAL: NCT00640939
Title: A Randomized, Double-Blind, Placebo-Controlled Study of the Efficacy and Safety of a Diclofenac Sodium Patch for the Topical Treatment of Pain Due to Mild to Moderate Tendonitis or Bursitis
Brief Title: Diclofenac Patch for Treatment of Mild to Moderate Tendonitis or Bursitis
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Cerimon Pharmaceuticals (Industry)
Collaborators: PPD Development, LP (Industry)
Responsible Party: Dan Levitt, MD, Cerimon Pharmaceuticals, Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DCF-003
Record Dates: First submitted 2008-03-18; First posted 2008-03-21 (Estimated); Last update posted 2008-08-06 (Estimated); Status verified 2008-08

CONDITIONS: Rotator Cuff Tendonitis; Bicipital Tendonitis; Subdeltoid Bursitis of the Shoulder; Subacromial Bursitis of the Shoulder; Medial Epicondylitis of the Elbow; Lateral Epicondylitis of the Elbow; DeQuervain's Tenosynovitis of the Wrist
Keywords: Tendonitis; Bursitis
MeSH Terms: conditions — Rotator Cuff Injuries; Tendinopathy; Bursitis | interventions — Diclofenac

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Active Comparator): Topical diclofenac sodium patch
  Interventions: Drug: diclofenac sodium
- B (Placebo Comparator): Topical patch identical in appearance to active comparator
  Interventions: Drug: Matching Placebo

INTERVENTIONS:
Drug: diclofenac sodium — 15 mg (1%) topical patch; measuring 7 cm by 10 cm; applied once daily
  Other Names: diclofenac
  Arms: A
Drug: Matching Placebo — Matching placebo patch, containing identical constituents to active patch except for diclofenac sodium; measuring 7 cm by 10 cm; applied once daily
  Other Names: placebo
  Arms: B

SUMMARY:
The primary purpose of this study is to assess the effectiveness of once daily application of a diclofenac sodium patch to the skin near or over the painful area. In this study, the location being studied will be one of the following: the affected shoulder, elbow, or wrist.

The secondary purpose of this study is to assess the safety and tolerability of the diclofenac patch on the subject's skin, in the location being studied.

DETAILED DESCRIPTION:
Cerimon Pharmaceuticals is investigating a topical patch formulation of diclofenac sodium containing 15 mg of diclofenac sodium for the local treatment of acute musculoskeletal pain.

ELIGIBILITY:
Inclusion Criteria:

* 18 years to 75 years of age
* Onset of painful upper extremity tendonitis or bursitis, no more than 21 days prior to study entry
* Eligible diagnoses are rotator cuff tendonitis, bicipital tendonitis or subdeltoid/subacromial bursitis of the shoulder, medial or lateral epicondylitis of the elbow, and DeQuervain's tenosynovitis of the wrist
* Spontaneous pain with motion or resisted motion and tenderness to palpation over the involved tendon(s), bursa, or epicondyle
* Presence of pain of at least 5, with a maximum of 9, on an 11-point Numerical Rating Scale (NRS)

Exclusion Criteria:

* Aspirin, or short half-life NSAID use within 12 hours, or longer half-life NSAID use within 24 hours prior to study entry (see Appendix B: for table of NSAIDs)
* Opioid use within 3 days prior to study entry
* Topical treatment, other than local ice or heat, applied to the painful region within 3 days prior to study entry
* History of peptic ulcer disease within 1 year prior to study entry, any history of gastrointestinal bleeding, or coagulation disorder
* A history of, or evidence for underlying articular disease such as osteoarthritis, rheumatoid arthritis, gout, or pseudogout (calcium pyrophosphate deposition disease)
* Clinically significant and poorly controlled pulmonary, gastrointestinal, hepatic, renal, endocrine, or cardiovascular disease
* A history of hypersensitivity to diclofenac or diclofenac-containing products
* A history of intolerance to acetaminophen (rescue medication in this trial)
* A history of skin sensitivity to adhesives (e.g. adhesive tape)
* Pregnant or breastfeeding women and women of child-bearing potential not using effective means of contraception

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 308 (Actual)
Dates: Start 2007-12; Primary Completion 2008-04 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Assess the efficacy of diclofenac in subjects with tendonitis or bursitis of the shoulder, elbow, or wrist. | 14 days

SECONDARY OUTCOMES:
Assess the safety and tolerability of diclofenac in subjects with tendonitis or bursitis of the shoulder, elbow, or wrist. | 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Dan Levitt, MD, Study Director — Cerimon Pharmaceuticals
Locations (1):
- PPD, Austin, Texas, United States